CLINICAL TRIAL: NCT04081038
Title: Dental Hygienists and Dentists as Providers of Oral Mucosa Screening and Brush Biopsies of Mucosal Lesions and Automated Artificial Intelligence Analysis of Cytology
Brief Title: Dental Hygienists and Dentists as Providers of Oral Mucosa Screening and Brush Biopsies
Acronym: mouthcancer
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Kristina Edman, Principal Investigator, Dalarna County Council, Sweden
Other Study IDs: Oral cancer screening
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Oral Cancer
Keywords: oral cancer screening
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Brush samples will be performed and the lesions obtained, analyzed for hrHPV and the presence of malignant cells or malignant associated cells.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Brush biopsy — Brush biopsy will be performed by dentists and dental hygienists

SUMMARY:
In 2007, The World Health Assembly (WHA) adopted a resolution to prevent oral cancer. The resolution urged the member states to ensure that measures against oral cancer was integrated into a national cancer control program by engaging and train dental personnel in screening, early diagnosis and treatment. Oral cancer is a severe oral health issue as it is potentially fatal and is the 5-6 most common tumor with approximately 275,000 cases for oral and 130,300 cases for pharyngeal cancers, excluding nasopharynx, globally. In Sweden,1000 new cases yearly is discovered and it is increasing. The explanation is an aging population and an increase in tonsil and tongue cancers caused by HPV, especially in younger subjects. This is due to changing sexual habits. Tumors caused by tobacco and alcohol are constant. Despite the decreasing prevalence of smoking and certain smoking-associated cancers, an increased incidence of tonsillar cancer has been seen in both Finland and Sweden. High risk HPV (hrHPV) oral cancer is also increasing.

DETAILED DESCRIPTION:
The 5 year survival of oral cancer in Sweden is 55 % and only 3-4% in advanced cases, with poor quality of life. The etiology is hrHPV, exposure to tobacco and alcohol in 65% and poor dental status. All are lifestyle factors so there are many opportunities for prevention and intervention. In 2016, 352 individuals in Sweden died in oral cancer compared with 135 individuals who died of cervical cancer. Leukoplakia (LP), erythroplakia (EP) and oral lichen planus (OLP) are the dominating oral premalignant entities. The diagnosis are clinical and often by biopsies. There are two types of leukoplakia, homogeneous and non-homogeneous. The nonhomogeneous have a risk of malignant transformation of 3.6-8.9% in Scandinavia. OLP is a chronic inflammatory lesion where the atrophic and erosive types have a risk of cancer development of 0.5-2%. The potential for prevention is high, as the risk factors are well known. The Clinical examination discloses any potentially malignant lesions. Screening for cervical cancer using brush sampling is a well-established method but for the early detection of oral premalignant and malignant lesions, this is not yet an accepted standard procedure. However, there are studies that clearly show that brush sampling is a reliable and safe method to identify oral cancer and their potentially malignant precursor. In subjects with suspected pre-malignant tissue changes, measures should be taken to organize to establish a diagnosis. The brush sampling technique are shown to be a faster less costly, and for the patient less troublesome technique than traditional incisional biopsies but both methods require today, referral to specialist care. Dental hygienists and dentists can most probably be trained to perform brush biopsies of oral premalignant lesions, and when diagnosed, the patient can be referred to a specialist to have the lesion excised, and required controls can possibly be carried out in the primary care. Dental health professionals have a responsibility to perform routine intra- and extraoral examination on their patients for detecting abnormalities. As dental hygienists and dentists often see their patients on a regular basis, they have the opportunity to provide this screening, and at an early stage detect abnormalities. In Sweden, education and training in examination of the oral mucosa is a part of the curriculum in dental hygienist education, so there is an expectation that the dental hygienist routinely perform tactile and visual examinations in practice. However, dental hygienists are not allowed to diagnose an oral mucosal lesion, but are trained to identify abnormalities and determine whether the patient needs referral to a dentist. It is also to expect that the dental hygienist and dentist are capable to identify risk behaviors, and recommend, and offer smoking cessation or refer the patient to a certified profession for smoking cessation. Being aware of the increasing number of head, neck, and oral tumors we need to focus on establishing easy, fast and affordable methods for diagnosis, managed at the general dental health clinics, preferably by dental hygienists and dentists.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Understand Swedish

Exclusion Criteria:

* Under 18 years of age
* Not understanding the Swedish language
* Previously mouth cancer diagnose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting Public Dental Health for routine check-ups.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Brush biopsy | 1 year
  Presence of tumor markers and hrHPV in premalignant oral lesions. Each item is scored 0 (no tumor markers) and 1 (tumor markers)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Gunnars Hellgren, Study Chair — Public Dental Health Region Dalarna
Locations (2):
- Sweden (2):
  - Kristina Edman, Falun, Dalarna County
  - Public Dental Service, Falun, Dalarna County

IPD SHARING:
Plan to Share IPD: Undecided